CLINICAL TRIAL: NCT03119467
Title: A Phase I/Ib, Study to Evaluate Safety and Efficacy of RP4010, in Patients With Relapsed or Refractory Lymphomas
Brief Title: Safety and Efficacy Study of RP4010, in Patients With Relapsed or Refractory Lymphomas
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study has been stopped after reviewing PK and safety results
Sponsor: Rhizen Pharmaceuticals SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RP4010-1601
Record Dates: First submitted 2017-04-10; First posted 2017-04-18 (Actual); Last update posted 2019-12-27 (Actual); Status verified 2019-12

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — RP4010

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): RP4010 to be administered
  Interventions: Drug: RP4010

INTERVENTIONS:
Drug: RP4010 — Escalating doses starting at 25 mg

SUMMARY:
A Phase I/Ib, Study to Evaluate Safety and Efficacy of RP4010, in Patients with Relapsed or Refractory Lymphomas

DETAILED DESCRIPTION:
Safety: Treatment-Emergent Adverse Events (AE); Treatment related AE, Serious Adverse Events (SAE) and Clinical significant AE; Dose Limiting Toxicities (DLT).

Pharmacokinetics (PK): Peak Plasma Concentration (Cmax), Area under the plasma concentration versus time curve (AUC), Time of Maximum Concentration Observed (Tmax).

Efficacy: Overall Response Rate (ORR), Progression Free Survival (PFS); Overall Survival (OS) and duration of Response (DoR).

ELIGIBILITY:
Inclusion Criteria:

* Refractory to or relapsed after at least 1 prior treatment line.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2
* Patients must be ≥18 years of age
* Able to give a written informed consent.

Exclusion Criteria:

* Patients receiving cancer therapy within 3 weeks prior to Cycle1 Day1 (C1D1).
* Patients with active Hepatitis B virus (HBV), Hepatitis C virus (HCV) or Human immune deficiency virus (HIV) infection
* Patients who received Allo-Stem cell Transplantation(Allo-SCT) within 12 months.
* Patients with graft versus-host disease (GVHD)
* Subjects who have received drugs that directly or indirectly inhibit calcineurin or Nuclear Factor of activated T cells (NFAT) activity .
* Patient with symptomatic, or history of documented congestive heart failure (NY Heart Association functional classification III-IV);
* Patient with Frederica's (QTcF) formulas (QTcF) ≥450 msec;
* Patient with angina not well-controlled by medication;
* Women who are pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-05-11 (Actual); Primary Completion 2019-11-29 (Actual); Study Completion 2019-12-19 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) Determination | 28 days
  To determine the maximum tolerated dose of RP4010 in patients with Relapsed or Refractory Non-Hodgkin Lymphoma

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax). | 24 hrs
  To assess the Maximum Plasma Concentration (Cmax).
Area under the curve (AUC) | 24 hrs
  To assess the Area under the plasma concentration versus time curve (AUC)
Anti-tumor activity-Overall response rate (ORR) | 2 months
  To assess the anti-tumor activity of RP4010 as determined by overall response rate (ORR)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (7):
  - University of Alabama, Birmingham, Alabama
  - City of Hope, Duarte, California
  - University of Colorado, Aurora, Colorado
  - University of Michigan, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Utah Cancer Specialists, Salt Lake City, Utah
- Australia (4):
  - St Vincent's Hospital, Sydney, New South Wales
  - Pindara Private Hospital, Benowa, Queensland
  - Brisbane Clinic for Lymphoma, Myeloma and Leukaemia, Greenslopes, Queensland
  - Epworth HealthCare, Richmond, Victoria

IPD SHARING:
Plan to Share IPD: Undecided